CLINICAL TRIAL: NCT06922370
Title: The Osteoarticular Manifestations in Patients With Gitelman Syndrome
Acronym: CPPD and more
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0670
Record Dates: First submitted 2025-04-03; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-03

CONDITIONS: Gitelman Syndrome; CPPD - Calcium Pyrophosphate Deposition Disease
MeSH Terms: conditions — Gitelman Syndrome; Chondrocalcinosis | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Gitelman Syndrome: Patients with clinically and genetically confirmed Gitelman syndrome.
  Interventions: Diagnostic Test: conventional radiograph or computed tomography

INTERVENTIONS:
Diagnostic Test: conventional radiograph or computed tomography — patients with gitelman syndrome evaluated with conventional radiograph or computed tomography

SUMMARY:
Patients with clinically and genetically confirmed Gitelman Syndrome are screened for CPPD, and the clinical and radiographic manifestations are collected and analyzed.

DETAILED DESCRIPTION:
Patients with clinically and genetically confirmed Gitelman Syndrome are screened for calcium pyrophosphate deposition, and the clinical data and radiographic manifestations are collected and analyzed to investigate the osteoarticular features in patients with Gitelman Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients confirmed with Gitelman Syndrome

Exclusion Criteria:

* Patients with other confounding situations such as Bartter Syndrome, hyperparathyroidism

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients clinically and genetically confirmed with Gitelman Syndrome
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
The presence of chondrocalcinosis | From the enrollment to the performance of the CPPD screen
  The presence of chondrocalcinosis on conventional radiograph or computed tomography in patients with Gitelman Syndrome

CONTACTS AND LOCATIONS:
Locations (1):
- the second affiliated hospital, Zhejiang University School of medicine, Hangzhou, Zhejiang, China